CLINICAL TRIAL: NCT05034133
Title: Durvalumab With Chemotherapy Followed by Sequential Radiotherapy for Limited Stage Small Cell Lung Cancer: A Single-arm Phase II Trial.
Brief Title: Durvalumab With Chemotherapy Followed by Sequential Radiotherapy for Limited Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Yuqing Huang, Director, Beijing Haidian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHHMEC-XM-2021-43
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Limited Stage Small Cell Lung Cancer
Keywords: Limited Stage Small Cell Lung Cancer; Durvalumab
MeSH Terms: interventions — durvalumab; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Patients with limited stage small cell lung cancer receive durvalumab with chemotherapy (Etoposide and Cisplatin) for receive 6 cycles, and then receive thoracic radiotherapy.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab (IV 1000mg on day 1) with chemotherapy (Etoposide and Cisplatin) for 6 cycles
  Other Names: Etoposide and Cisplatin

SUMMARY:
This is a single arm Phase II study, in which 6 cycles of durvalumab with chemotherapy (Etoposide and Cisplatin) and durvalumab followed by Sequential radiotherapy for limited stage small cell lung cancer.

DETAILED DESCRIPTION:
Primary Outcome Measures:

Progression free survival

Secondary Outcome Measures:

Overall survival Safety analysis

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Histologically confirmed small cell lung cancer
3. Limited disease, defined as disease confined to one hemithorax, the mediastinum, and the bilateral supraclavicular fossae.
4. Age > 18 years at time of study entry
5. ECOG performance status of 0 to 1
6. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC ≥ 1.5 (or 1.0) x (> 1500 per mm3)
   * Platelet count ≥ 100 (or 75) x 109/L (>75,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and

   Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males: Creatinine CL (mL/min) =Weight (kg) x (140 - Age)/ 72 x serum creatinine (mg/dL) Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85/ 72 x serum creatinine (mg/dL)
7. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
8. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Patients with extensive disease small-cell lung cancer
3. Patients who previously received radiotherapy to the thorax or chemotherapy for small cell lung cancer
4. Participation in another clinical study with an investigational product at any time
5. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
7. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogenic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
11. Uncontrolled illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
    * Adequately treated early gastric cancer
13. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
14. History of active primary immunodeficiency
15. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
    * Steroids as antiemetics for 5FU/cisplatin chemotherapy
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
21. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  The PFS time is defined as time from enrollment to locoregional or systemic

SECONDARY OUTCOMES:
OS（Overall Survival） | From enrollment until death (up to 24 months)
  OS was defined as time from date of enrollment to date of death due to any cause.
Safety analysis | 1 year
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Huang, Director, Study Director — Beijing Haidian Hospital
Locations (1):
- Beijing Haidian Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No